CLINICAL TRIAL: NCT03201679
Title: The Association Between Preoperative Sepsis and the Mortality After Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Sara Tantholdt-Hansen, Medical student, Bispebjerg Hospital
Other Study IDs: Preoperative sepsis 2017
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Sepsis; Hip Fractures
Keywords: SIRS, systemic inflammatory response syndrome; Hip Fracture Surgery; Sepsis; Mortality
MeSH Terms: conditions — Sepsis; Hip Fractures; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with preoperative sepsis: Sepsis defined as SIRS plus a positive culture from any site.
  Interventions: Procedure: Repair of hip fracture
- Patients without preoperative sepsis
  Interventions: Procedure: Repair of hip fracture

INTERVENTIONS:
Procedure: Repair of hip fracture — Patients undergoing hip fracture surgery

SUMMARY:
The worldwide occurrence of hip fracture is high with an annual incidence of approximately 100 per 100.000 people. Mortality for patients undergoing hip fracture surgery is high with a 30-day mortality rate varying between 4.5 and 13.3 %. It is agreed that non-modifiable factors such as age, gender and pre-existing comorbidities contribute to early death of hip fracture patients. However, not many studies have focused on preoperative sepsis as a potential risk factor. Hip fracture patients are commonly identified with sepsis after surgery, but the extent of preoperative sepsis and its consequences are sparsely elucidated. Being able to identify patients at higher risk of postoperative mortality could potentially improve outcome and extensive hospital registries of vital signs and cultures allow identification of preoperative sepsis.

The aim of this study is to assess the association between preoperative sepsis and the 30-day mortality after hip fracture surgery.

DETAILED DESCRIPTION:
This study will be a retrospective analysis of a set of data collected prospectively. Data on relevant cultures, blood samples, co-morbidities, time to surgery and 30-day mortality will be extracted from patient records and clinical databases to examine the pre- and postoperative status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following ICD-10 diagnoses for hip fracture: DS720(Fracture of neck of femur), DS721 (Pertrochanteric fracture), DS721A(Intertrochanteric fracture), DS721B (Trochanteric fracture), DS722 (Subtrochanteric fracture)
* Patients who underwent surgery for hip fracture.
* Age > 18 years

Exclusion Criteria:

* Patients with a pathologic hip fracture related to an underlying metastatic disease (ICD-10: DM907).
* Patients with incomplete preoperative data. All patients must have at least one record of each of the following variables within 72 hours prior to hip fracture surgery: temperature, heartrate, respiratory rate and blood leukocytes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients admitted with a primary diagnosis of hip fracture and who underwent hip fracture surgery between January 1, 2014 and December 31, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 1967 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

SECONDARY OUTCOMES:
Admission to intensive care | 30 days
  yes/no
Length of hospital stay | 30 days
  in days

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, PhD, Study Chair — Department of Aneasthesia and Intensive Care, Bispebjerg Hospital

REFERENCES:
- [Background] Smith T, Pelpola K, Ball M, Ong A, Myint PK. Pre-operative indicators for mortality following hip fracture surgery: a systematic review and meta-analysis. Age Ageing. 2014 Jul;43(4):464-71. doi: 10.1093/ageing/afu065. Epub 2014 Jun 3. PMID 24895018
- [Background] Khan MA, Hossain FS, Ahmed I, Muthukumar N, Mohsen A. Predictors of early mortality after hip fracture surgery. Int Orthop. 2013 Nov;37(11):2119-24. doi: 10.1007/s00264-013-2068-1. Epub 2013 Aug 28. PMID 23982637
- [Background] Deakin DE, Boulton C, Moran CG. Mortality and causes of death among patients with isolated limb and pelvic fractures. Injury. 2007 Mar;38(3):312-7. doi: 10.1016/j.injury.2006.09.024. Epub 2006 Dec 4. PMID 17141780
- [Background] Hu F, Jiang C, Shen J, Tang P, Wang Y. Preoperative predictors for mortality following hip fracture surgery: a systematic review and meta-analysis. Injury. 2012 Jun;43(6):676-85. doi: 10.1016/j.injury.2011.05.017. Epub 2011 Jun 17. PMID 21683355
- [Background] Pedersen NE, Rasmussen LS, Petersen JA, Gerds TA, Ostergaard D, Lippert A. A critical assessment of early warning score records in 168,000 patients. J Clin Monit Comput. 2018 Feb;32(1):109-116. doi: 10.1007/s10877-017-0003-5. Epub 2017 Feb 25. PMID 28238106